CLINICAL TRIAL: NCT04240158
Title: Evaluating the Safety, Tolerability, and Pharmacodynamic Properties of IW-6463 in Healthy Elderly Subjects
Brief Title: IW-6463 Safety Study in Healthy Elderly Subjects
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Some subjects could not complete the second crossover period due to COVID-19-related site closure. The study was closed to allow analysis of all collected data.
Sponsor: Tisento Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: C6463-102; CY6463 (Other: Cyclerion Therapeutics)
Record Dates: First submitted 2020-01-21; First posted 2020-01-27 (Actual); Last update posted 2024-08-16 (Actual); Status verified 2024-08

CONDITIONS: Other

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- IW-6463 (Experimental): IW-6463 tablets administered orally
  Interventions: Drug: IW-6463
- Placebo (Placebo Comparator): Matching placebo tablets administered orally
  Interventions: Drug: Matching Placebo

INTERVENTIONS:
Drug: IW-6463 — IW-6463 Tablet
  Other Names: CY6463; zagociguat
  Arms: IW-6463
Drug: Matching Placebo — Matching Placebo Tablet
  Arms: Placebo

SUMMARY:
This is a randomized, double-blind, placebo-controlled, 2-way cross-over study in healthy male and female elderly participants.

DETAILED DESCRIPTION:
Participants will receive up to a total of 30 daily doses of study drug (15 days of daily IW-6463, only; 15 days of daily placebo, only) administered across two 15-day dosing periods (Period 1 and Period 2). The dosing periods will be separated by a 27-day washout. Participants will be randomized to a sequence of receiving IW-6463 for Period 1 and then placebo for Period 2, or vice versa.

ELIGIBILITY:
Inclusion Criteria:

* Subject is an ambulatory adult at least 65 years old at the screening visit
* Subject is in good health and has no clinically significant findings on physical examination
* Female participants must be postmenopausal. A postmenopausal state is defined as no menses for ≥12 consecutive months without an alternative medical cause. A high follicle-stimulating hormone (FSH) level at screening (>40 IU/L or mIU/mL) in the postmenopausal range may be used to confirm a postmenopausal state.
* Male participants who have not been surgically sterilized by vasectomy (conducted ≥60 days before the Screening Visit or confirmed via sperm analysis) must agree contraceptive use per protocol
* Men must also agree to not donate sperm throughout the study and for 3 months after the final dose of study drug
* Other inclusion criteria per protocol

Exclusion Criteria:

* Any active or unstable clinically significant medical condition
* Other exclusion criteria per protocol

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 24 (Actual)
Dates: Start 2020-01-06 (Actual); Primary Completion 2020-05-22 (Actual); Study Completion 2020-05-22 (Actual)

PRIMARY OUTCOMES:
Change From Baseline in Cerebral Blood Flow (CBF) at Day 15 | Baseline, 15 days
  Change from baseline in CBF as measured by magnetic resonance imaging (MRI) and arterial spin labeling (ASL) after administration of IW-6463 vs. placebo
Number of Participants With ≥1 Treatment-Emergent Adverse Events (TEAEs) | Up to 42 days

CONTACTS AND LOCATIONS:
Overall Officials: Chad Glasser, PharmD, Study Director — Cyclerion Therapeutics, Inc; Geert Jan Groeneveld, MSc, Principal Investigator — Centre for Human Drug Research
Locations (1):
- Centre for Human Drug Research (CHDR), Leiden, Netherlands

IPD SHARING:
Plan to Share IPD: No